CLINICAL TRIAL: NCT06190483
Title: Effect of Benzodiazepine on Corticolimbic Activation, GABA and Glutamate in Subjects at Clinical High Risk of Psychosis
Brief Title: Investigating the Role of Diazepam on Brain Function and Chemistry in Psychosis Risk
Acronym: BENZOGAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Wellcome Trust (Other); The Royal Society (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 18/LO/0618
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Prodromal Schizophrenia
MeSH Terms: conditions — Schizotypal Personality Disorder | interventions — Diazepam; Tablets; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diazepam/Placebo (Experimental): Participant's receive diazepam on 1st MRI scan, and placebo (ascorbic acid) on 2nd MRI scan
  Interventions: Drug: Diazepam 5 Mg Oral Tablet; Drug: Ascorbic Acid 50 Mg Oral Tablet
- Placebo/Diazepam (Experimental): Participant's receive placebo (ascorbic acid) on 1st MRI scan, and diazepam on 2nd MRI scan
  Interventions: Drug: Diazepam 5 Mg Oral Tablet; Drug: Ascorbic Acid 50 Mg Oral Tablet

INTERVENTIONS:
Drug: Diazepam 5 Mg Oral Tablet — Single dose given orally (opaque capsule) 60 minutes prior to MRI scan
  Other Names: Diazepam
Drug: Ascorbic Acid 50 Mg Oral Tablet — Single dose given orally (opaque capsule) 60 minutes prior to MRI scan
  Other Names: Placebo

SUMMARY:
This study will investigate whether a single dose of diazepam (5mg) compared to placebo can modulate brain chemistry (GABA/glutamate levels) and function (blood flow, neural response and connectivity during tasks and at-rest) in 24 individuals at clinical high-risk for psychosis.

DETAILED DESCRIPTION:
The pathophysiology of psychosis involves elevated subcortical dopamine function, but the factors driving this are still unclear. Evidence from a neurodevelopmental animal model of psychosis suggests that this arises through a pathway linking psychosocial stress, corticolimbic hyperresponsivity, and GABA/glutamate imbalance. In response to stress/negative emotion, amygdala hyperresponsivity decreases GABA interneuron function in the hippocampus through strong direct projections. Decreased hippocampal GABA function leads to disinhibition of hippocampal pyramidal cells, elevating local activity and glutamate levels. Increased output from the hippocampus to the striatum elevates dopamine release in the striatum, and increases the firing of dopaminergic neurons in the midbrain. These neurobiological effects are associated with cognitive (e.g., working memory) and emotional deficits (e.g., increased anxiety). Moreover, peripubertal (premorbid) administration of benzodiazepines at anxiolytic doses to this animal of psychosis is shown to normalise hippocampal activity, thereby preventing the emergence of striatal hyperdopaminergia and associated behavioural abnormalities in adulthood. Collectively, these findings indicate that GABA dysfunction and emotional hyperresponsivity may play a critical role in the development of psychosis in humans, and suggest that clinical interventions targeting this pathway have the potential to reduce the risk of developing the disorder.

This study will use multimodal neuroimaging (MRS, ASL, rs-fMRI, tb-fMRI) to assess whether the acute administration of a benzodiazepine can modulate the pathway linking corticolimbic response and GABA/glutamate levels in people in the premorbid stage of psychosis (at "clinical high risk", CHR). Using a randomised, double-blind, placebo-controlled, crossover design, 24 CHR-P participants will undergo two MRI sessions, once under an acute oral dose of diazepam (5 mg; generic) and once under oral placebo (50 mg ascorbic acid), with a minimum 3-week washout period between visits.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-40 years
* Capacity to consent to participation in the study
* Inclusion into one of three groups as assessed by the CAARMS: i) genetic vulnerability group, ii) attenuated psychosis group, iii) brief intermittent psychosis symptoms group. This instrument has been modified to additionally allow the scoring of the SIPS v.520. The scoring of the SIPS v.5 is included for comparative purposes and does not constitute inclusion criteria.
* Inclusion based on meeting criteria for "basic symptoms" which are assessed using the Schizophrenia Proneness Instrument (SPI-A)21

Exclusion Criteria:

* History of neurological disorders
* Current exposure to any drug with potential GABAergic or glutamatergic effects other than antipsychotics, mood stabilisers, antidepressants. This includes opiates, psychostimulants, benzodiazepines, atomoxetine, memantine, ketamine, cough medication containing dextromethorphan
* Current or past exposure to any antipsychotic medication
* Pregnancy/breastfeeding
* Contra-indication to MRI scanning (e.g., metal in body, such as pacemakers or implants, claustrophobia)
* IQ < 70 as determined with the shortened version of the Wechsler Adult Intelligence Scale III (WAIS-III)22

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
GABA/Glutamate concentrations (Magnetic Resonance Spectroscopy) | Assessed at 1st and 2nd MRI scan (~2 and ~6 weeks, respectively, after enrolment)
  To evaluate the acute effect of a benzodiazepine drug (diazepam) on GABA and glutamate concentrations in people at clinical high risk of psychosis (CHR).

SECONDARY OUTCOMES:
Cerebral blood flow (Arterial Spin Labelling) | Assessed at 1st and 2nd MRI scan (~2 and ~6 weeks, respectively, after enrolment)
  To determine if hippocampal cerebral blood flow is normalised in subjects at CHR under the diazepam condition compared to placebo
Functional connectivity (Resting State Functional Magnetic Resonance Imaging) | Assessed at 1st and 2nd MRI scan (~2 and ~6 weeks, respectively, after enrolment)
  To determine if hippocampal resting functional connectivity is normalised in subjects at CHR under the diazepam condition compared to placebo
Neural response to emotional stimuli (Task Based Functional Magnetic Resonance Imaging) | Assessed at 1st and 2nd MRI scan (~2 and ~6 weeks, respectively, after enrolment)
  To determine if neural response to emotional stimuli and during working memory is normalised in subjects at CHR under the diazepam condition compared to placebo
Neural response during working memory (Task Based Functional Magnetic Resonance Imaging) | Assessed at 1st and 2nd MRI scan (~2 and ~6 weeks, respectively, after enrolment)
  To determine if neural response during working memory is normalised in subjects at CHR under the diazepam condition compared to placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Psychiatry, Psychology and Neuroscience, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No